CLINICAL TRIAL: NCT00477074
Title: Pulmonary and Systemic Hepatocyte Anb Keratinocyte Growth Factors in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Pulmonary and Systemic Hepatocyte Growth Factors in Patients With COPD
Status: Completed | Type: Observational
Sponsor: Hospital Universitari Son Dureta (Other)
Collaborators: Sociedad Española de Neumología y Cirugía Torácica (Other); Fundacion Caubet-Cimera Islas Baleares (Other)
Other Study IDs: SEPAR2002FG
Record Dates: First submitted 2007-05-18; First posted 2007-05-22 (Estimated); Last update posted 2007-05-22 (Estimated); Status verified 2007-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive pulmonary disease; emphysema; inflammation; repair
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Inflammation | interventions — Bronchoalveolar Lavage; Hematologic Tests

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: bronchoalveolar lavage, blood analysis

SUMMARY:
The role of HGF and KGF in COPD is poorly known. Plantier et al found that cultured fibroblasts harvested from patients with emphysema produced less HGF (but similar amounts of KGF) than controls, and Bonay et al found a direct relationship between the severity of airflow obstruction and HGF mRNA content in lung samples of smokers. These two studies suggest, therefore, that the pulmonary regulation of HGF may be abnormal in patients with COPD. However, both HGF and KGF can also be released by extra-pulmonary organs, thus having the potential to act systemically. Given the current clinical relevance attributed to the systemic effects of COPD, in this study we compared the levels of HGF and KGF in the pulmonary (bronchoalveolar lavage (BAL) fluid) and systemic compartment (circulating blood) of smokers with and without COPD and never smokers.

DETAILED DESCRIPTION:
Background: The potential role of growth factors in COPD has begun to be addressed only recently and is still poorly understood. In this study we investigate potential abnormalities of hepatocyte growth factor (HGF) and keratinocyte growth factor (KGF) in patients with COPD.

Methods: To this end, we compared the levels of HGF and KGF, measured by ELISA, in bronchoalveolar lavage (BAL) fluid and in serum in 18 patients with COPD (62 ± 2 yrs, FEV1 57 ± 4% ref, X ± SEM), 18 smokers with normal lung function (58 ± 2 yrs., FEV1 90 ± 4% ref) and 8 never smokers (67 ± 7 yrs, 94 ± 4% ref).

Results: We found that, in BAL, HGF levels were higher in patients with COPD than in the other two groups whereas, in serum, HGF concentration was highest in smokers with normal lung function (p<0.01). KGF levels were not significantly different between groups, neither in blood nor in BAL, (most values were below the detection limit).

Conclusions: These results highlight a different response of HGF in BAL and serum in smokers with and without COPD that may be relevant for tissue repair in COPD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with COPD (GOLD II-III) 1, smokers without chronic bronchitis or dyspnea and with normal lung function, and never smokers who required bronchoscopy for clinical purposes.

Exclusion Criteria:

* Acute exacerbation last three months
* Chronic lung diseases (asthma, bronchiectasis and interstitial lung diseases) and cardiac, hepatic or renal failure.
* Systemic steroid treatment

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2004-01; Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaume Sauleda, Principal Investigator — Hospital Universitari Son Dureta
Locations (1):
- Servei Pneumologia. Hospital Universitari Son Dureta, Palma de Mallorca, Balearic Islands, Spain

REFERENCES:
- [Background] Bonay M, Boutten A, Lecon-Malas V, Marchal J, Soler P, Fournier M, Leseche G, Dehoux M, Crestani B. Hepatocyte and keratinocyte growth factors and their receptors in human lung emphysema. BMC Pulm Med. 2005 Oct 10;5:13. doi: 10.1186/1471-2466-5-13. PMID 16216128
- [Background] Sugahara K, Matsumoto M, Baba T, Nakamura T, Kawamoto T. Elevation of serum human hepatocyte growth factor (HGF) level in patients with pneumonectomy during a perioperative period. Intensive Care Med. 1998 May;24(5):434-7. doi: 10.1007/s001340050592. PMID 9660257
- [Background] Shigemura N, Sawa Y, Mizuno S, Ono M, Minami M, Okumura M, Nakamura T, Kaneda Y, Matsuda H. Induction of compensatory lung growth in pulmonary emphysema improves surgical outcomes in rats. Am J Respir Crit Care Med. 2005 Jun 1;171(11):1237-45. doi: 10.1164/rccm.200411-1518OC. Epub 2005 Mar 11. PMID 15764723
- [Background] Plantier L, Marchand-Adam S, Marchal-Somme J, Leseche G, Fournier M, Dehoux M, Aubier M, Crestani B. Defect of hepatocyte growth factor production by fibroblasts in human pulmonary emphysema. Am J Physiol Lung Cell Mol Physiol. 2005 Apr;288(4):L641-7. doi: 10.1152/ajplung.00249.2004. Epub 2004 Dec 3. PMID 15579628
- [Background] Mason RJ. Hepatocyte growth factor: the key to alveolar septation? Am J Respir Cell Mol Biol. 2002 May;26(5):517-20. doi: 10.1165/ajrcmb.26.5.f239. No abstract available. PMID 11970901
- [Background] Stern JB, Fierobe L, Paugam C, Rolland C, Dehoux M, Petiet A, Dombret MC, Mantz J, Aubier M, Crestani B. Keratinocyte growth factor and hepatocyte growth factor in bronchoalveolar lavage fluid in acute respiratory distress syndrome patients. Crit Care Med. 2000 Jul;28(7):2326-33. doi: 10.1097/00003246-200007000-00024. PMID 10921560
- [Background] Welsh DA, Summer WR, Dobard EP, Nelson S, Mason CM. Keratinocyte growth factor prevents ventilator-induced lung injury in an ex vivo rat model. Am J Respir Crit Care Med. 2000 Sep;162(3 Pt 1):1081-6. doi: 10.1164/ajrccm.162.3.9908099. PMID 10988134
- See also: Spanish Respiratory Society — http://www.separ.es